CLINICAL TRIAL: NCT00449423
Title: Metabolic Modulation as Treatment in Acute Heart Failure
Acronym: MEMO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: due to slow recruitment
Sponsor: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20060810
Record Dates: First submitted 2007-03-19; First posted 2007-03-20 (Estimated); Last update posted 2007-10-25 (Estimated); Status verified 2007-10

CONDITIONS: Acute Heart Failure
Keywords: Acute heart failure; Metabolic modulation
MeSH Terms: interventions — acipimox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: acipimox

SUMMARY:
The primary objective of this study is to evaluate whether metabolic modulation improves hemodynamics and outcome in acute heart failure

DETAILED DESCRIPTION:
Acute heart failure is a serious disease that despite modern therapies carries a high mortality. Inotropic drugs improve patient status but yield a higher risk of death. Previous studies have shown that myocardial contractility improves when glucose fermentation is up regulated and decreases when Free Fatty Acids are high. In a placebo-controlled design we wish to shift myocardial substrate metabolism towards increased glucose uptake and utilization and measure hemodynamics and biochemical markers of metabolism and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Acute heart failure
* NYHA class III - IV.
* ejection fraction <35

Exclusion Criteria:

* Age <18 år or >85 år,
* allergy
* renal failure
* recently developed brady- or tachy-arrythmias
* Serious infection
* Heart failure due to restrictive or hypertrophic cardiomyopathy or stenotic valvular heart disease
* Recent Myocardial infarction (<6 Weeks)
* Pulmonary Wedge pressure >30 mm Hg
* diabetes mellitus treated with insulin
* peptic ulcer
* pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2007-03; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Cardiac index
pulmonary Wedge Pressure
Ejection fraction

SECONDARY OUTCOMES:
myocardial glucose- and Free Fatty Acid-extraction
cardiac output
Regional left ventricle function
outcome day 6 and 30

CONTACTS AND LOCATIONS:
Overall Officials: Mads Halbirk, dr., Principal Investigator — Aarhus University Hospital, Department of Cardiology
Locations (1):
- Aarhus University Hospital, Skejby Sygehus, Department of Cardiology, Aarhus, Aarhus, Denmark